CLINICAL TRIAL: NCT06196944
Title: Effects of Augmentative and Alternative Communication in Children With Cerebral Palsy
Brief Title: Effects of Augmentative and Alternative Communication in Children With Cerebral Palsy Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2723 Sibgha
Record Dates: First submitted 2023-10-26; First posted 2024-01-09 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Augmentative and Alternative Communication Devices; Speech and Language Therapy; Assisted Communication
MeSH Terms: conditions — Cerebral Palsy; Communication Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmentative Alternative Communication (Other): Traditional treatment
  Interventions: Behavioral: Augmentative Alternative Communication
- Augmentative Alternative Communication Device (Other): 3 sessions per week for 40 minutes
  Interventions: Other: Augmentative Alternative Communication Device

INTERVENTIONS:
Behavioral: Augmentative Alternative Communication — Traditional Method
  Arms: Augmentative Alternative Communication
Other: Augmentative Alternative Communication Device — Augmentative Alternative Communication Device 3 session for 40 minutes
  Arms: Augmentative Alternative Communication Device

SUMMARY:
Cerebral Palsy is a neuromuscular disorder that causes multiple disabilities in an individual.

Children's ability to rely on speech as a primary mode of communication can be compromised by cerebral palsy. Children with communication difficulties face many barriers to participating in everyday life and have a heightened risk of social isolation and mental health problems.

So, augmentative, and alternative communication (AAC) strategies and tools are helpful for children with CP. AAC is classified into manual signs and symbols, and low, mid, and high- tech communication aids form part of a total communication approach whereby all potential modalities of communication are explored and supported. The World Health Organization International Classification of Function, Disability, and Health for Children and Youth is increasingly being used to support decision-making. The study will be carried out at Rising Sun Institute for Special Children. The study design for this study is Randomized Control Trials. The convenience Sampling Technique will be used to collect data and 16 children with cerebral palsy will be included in this study. Both males and females with the age range of 3-15 years will be included in this study. The children will be randomly assigned into groups, group A will be allocated 8 children as the control group, and in group B, 8 as the treatment/ interventional group. Dysarthric Profile will be used for assessment purposes and aided Augmentative and Alternative communication system for the intervention. The pre-assessment of the child's Early Functional development will be done. Then, the low- tech (PECS) will be used for 6 weeks for the intervention. We will take 3 sessions per week for 40 minutes for the treatment group while the control group will remain the same. After the end of 6 weeks, the post-assessment of the child's Early Functional development will also be done. This indicates the effectiveness of AAC devices in the communication of children with Cerebral Palsy. The use of AAC methods could help to reduce aggressiveness among children with cerebral palsy. Moreover, AAC-based information and tools enable them to create environments that will support or enhance the ability of people with complex communication needs to interact with family members, peers, teachers, and others.

DETAILED DESCRIPTION:
Communication abilities are basic developmental skills within the adaptive development of a person, particularly during childhood. Therefore, children and teenagers with receptive and expressive communication impairment face challenges over numerous life spans. Several kinds of literature have detailed that they appear to have higher rates of psychosocial disabilities, lower scholarly performance, more peer rejection, and troubles in their social intelligence, compared to normal developing peers. Roughly 8% of children between the ages of 3 and 17 a long time within the United States face language and communication problems, and thus may need extra support for normal communication skills. (1) Individual with complex communication needs is likely to come from several different conditions (e.g., cerebral palsy).

Even though some individuals with these challenges will be effectively supported by assistance from other people, such as teachers, caregivers, community workers, and family friends, there will be some who are underserved due to the lack of rehabilitation specialists in low-income countries. (2) Cerebral Palsy has a neurogenic origin leading to physical impairment in children or may be caused by maternal (perinatal, natal, and postnatal injuries). The common types of cerebral palsy are spastic, flaccid, ataxic, or mixed types, determined by the site of the lesion in the brain. It adversely affects gross and fine motor development, receptive-expressive language skills, speech (articulation), voice (intensity, pitch, and quality), and fluency, depending on etiology. (3) The prevalence of CP in the United States ranges from 3-4 per 1000 live births.

Within the 2009-16 period, the prevalence of CP in children matured 3-17 a long time was 3.2 per 1000. The prevalence of low birth weight (LBW) and preterm in live births are altogether higher (40-100/1000). According to a study in Swabi, Pakistan, the prevalence of CP is 1.22 per 1000 live births. However, country-wide statistics are not found but 6.9% incidence of CP children admission in a Lahore hospital out of the 6.7% pediatric neurological admissions.

Research suggests evidence of the impact of the use of AAC-implemented intervention on 9 children in rural Kenya who have complex communication needs. The intervention used mainly low- tech materials that were specifically designed to strengthen the child's communication while remembering the caregiver's natural expertise. A pretest-posttest design was used in this study. Data were gathered using an adapted version of the Communication Profile, which was based on the International Classification of Functioning, Disability, and Health (ICF) framework. Qualitative analysis was conducted in the final section of the study. The data provided evidence of statistically significant positive changes in the communication of children with cerebral palsy at the levels of Body Structure Function and Activities. Also, the analysis revealed the positive perception of parents regarding AAC. (2) OBJECTIVE

To investigate the effects of Augmentative and Alternative Communication in Children with Cerebral Palsy. HYPOTHESES NULL HYPOTHESIS Ho= Augmentative and alternative communication is not an effective intervention for children with cerebral palsy.

ALTERNATE HYPOTHESIS H A =Augmentative and alternative communication is an effective intervention for children with cerebral palsy. STUDY DESIGN Randomized Control trials

SETTING Rising Sun Institute for Special Children

DURATION OF THE STUDY 6 months after the approval of the synopsis

SAMPLE SIZE This sample is 16 according to the literature review. STUDY GROUPS Group A: Treatment Group will consist of 8 children with cerebral palsy. Group B: Control Group will consist of 8 children with cerebral palsy.

SAMPLING TECHNIQUE Simple Random Sampling Technique

DATA COLLECTION TOOL Dysarthric Profile will be used for assessment purposes and a low-tech Picture Exchange Communication System (PECS) for the intervention.

DATA COLLECTION PROCEDURE:

According to the inclusion criteria, 16 children will be recruited. The children will be assigned into groups. The randomly selected groups will be allocated 8 children as the control group and 8 as the treatment/ interventional group. A pre-assessment of the child's Early Functional development will be done. After that, the low-tech intervention will be applied for 6 weeks (3 sessions per week for 40 minutes) to the treatment group while the control group will remain the same. After the end of 6 weeks, the post-assessment of the child's Early Functional development will be done. This indicates the effectiveness of AAC in the communication of children with Cerebral Palsy.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female children who have a confirmed diagnosis of cerebral palsy as reported in the medical history by a medical specialist (i.e., neurologist, pediatrician)

Exclusion Criteria:

* No child will be with any kind of comorbidity symptoms or any known additional disabilities (e.g., Down syndrome, autism spectrum disorder, seizure disorder, blindness, etc.)

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Dysarthric Profile | 16 weeks
  Dysarthria Rating Scale Rate speech by assigning a value of 0-4 to each of the dimensions listed below (0 = normal; 1 mild; 2 moderate; 3 marked; 4 severely deviant). A + should be used to indicate excessive or high; - should be used to indicate reduced or low when appropriate.
Picture Exchange Communication System (PECS) | 16 weeks
  The Picture Exchange Communication System (PECS) is a way for autistic people to communicate without relying on speech. To communicate, people use cards with pictures, symbols, words or photographs to ask for things, comment on things or answer questions.

CONTACTS AND LOCATIONS:
Overall Officials: Nazia Mumtaz, Principal Investigator — Riphah International University
Locations (1):
- Sibgha Shafique, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No